CLINICAL TRIAL: NCT05806060
Title: Precise Treatment for BLIS Subtype of Triple-negative Breast Cancer in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer
Brief Title: Precise Treatment for BLIS Subtype of TNBC in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer
Acronym: BCTOP-T-M01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-TNBC-BLIS
Record Dates: First submitted 2023-03-09; First posted 2023-04-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Capecitabine; Bevacizumab; eribulin; CCDC6 protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- De novo or DFI≥12m Arm 1 (Experimental): If patients were De novo or their disease-free interval (DFI) were more than or equal to 12 months and were randomized to experimental arm, they would receive VEGFR BP102 with nab-palitaxel (Nab-P). And maintained by VEGFR and capecitabine if intolerable toxicity was observed with no progression.
  Interventions: Drug: VEGFR and nab-paclitaxel, with maintenance of VEGFR and capecitabine
- De novo or DFI≥12m Arm 2 (Active Comparator): If patients were De novo or their disease-free interval (DFI) were more than or equal to 12 months and were randomized to control arm, they would receive nab-palitaxel (Nab-P). And maintained by capecitabine if intolerable toxicity was observed with no progression.
  Interventions: Drug: nab-paclitaxel, with maintenance of capecitabine
- DFI<12m Arm 1 (Experimental): If patients' disease-free interval (DFI) were less than 12 months and were randomized to experimental arm, they would receive VEGFR BP102 with treatment of physician's choice (TPC).
  Interventions: Drug: VEGFR and TPC
- DFI<12m Arm 2 (Active Comparator): If patients' disease-free interval (DFI) were less than 12 months and were randomized to control arm, they would receive physician's choice (TPC).
  Interventions: Drug: Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1

INTERVENTIONS:
Drug: VEGFR and nab-paclitaxel, with maintenance of VEGFR and capecitabine — VEGFR bevacizumab 10mg/kg d1,15 ivgtt + nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle. Capecitabine with bevacizumab maintenance if intolerable toxicity was observed with no progression. Capecitabine maintenance 1000mg/m2 po bid d1-d14 every 3 weeks and bevacizumab 10mg/kg d1,15 ivgtt every 4 weeks.
  Other Names: Bevacizumab (BP102)
  Arms: De novo or DFI≥12m Arm 1
Drug: nab-paclitaxel, with maintenance of capecitabine — Nab-paclitaxel 100mg/m2 d1,8,15 ivgtt, 4 weeks as a cycle. Capecitabine maintenance if intolerable toxicity was observed with no progression. Capecitabine maintenance 1000mg/m2 po bid d1-d14 every 3 weeks.
  Arms: De novo or DFI≥12m Arm 2
Drug: Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1 — TPC
  Arms: DFI<12m Arm 2
Drug: VEGFR and TPC — VEGFR bevacizumab and TPC
  Other Names: Bevacizumab (BP102)
  Arms: DFI<12m Arm 1

SUMMARY:
The study is being conducted to evaluate VEGFR BP102 with nab-paclitaxe or treatment of physician's choice (TPC) versus nab-paclitaxe or TPC in patients for basal-like immune suppressed (BLIS) subtype of triple-negative breast cancer (TNBC) in the first-line teatment of unresectable locally advanced or metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression) with BLIS subtype
* Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resection
* Patients had received no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer
* At least one measurable or non-measurable lesion according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), which didn't receive radiation therapy
* The functions of major organs are basically normal
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Have the cognitive ability to understand the protocol and be willing to participate and to be followed up

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Significant cardiovascular disease
* Adverse reactions of Grade ≥1 that are still continuing due to previous treatments. Exceptions are those of hair loss or which researchers take it as exception
* Major surgery was performed within 3 weeks of the first course of trial treatment (except for minor outpatient surgery, such as placement of vascular access)
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Other malignancies within 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, or skin squamous cell carcinoma
* Inability to swallow, chronic diarrhea and intestinal obstruction, there are multiple factors that affect the use and absorption of drugs
* Presence of third-space fluid accumulation that cannot be controlled by drainage or other methods (such as excessive pleural fluid and ascites)
* Participated in clinical trials of other antitumor drugs within 4 weeks before first taking the investigational drug
* Long-term unhealing wound or incomplete healing of fracture
* Patients with known active HBV or HCV infection or hepatitis B DNA≥500, or chronic phase with abnormal liver function
* Allergic constitution, or known allergic history of the drug components of this trial; Or allergic to other monoclonal antibodies
* Patients with a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding within the past 6 months, such as esophageal varicose veins with bleeding risk, locally active ulcer lesions, stool occult blood ≥ (++), were not allowed to enter the group; If there is occult blood in the stool (+), gastroscopy is required
* Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 28 days before participating in this trial
* Urine protein ≥2+ and 24h urine protein quantitative > 1.0 g
* Patients suffering from hypertension and unable to reach the normal range after antihypertensive drug treatment (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 1.5 years)
  time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
ORR | max 6 months
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
DoR | max 6 months
  Duration of Overall Response.The date of the first assessed PR/CR (according to RECIST 1.1) to the date of the first assessed tumor progression (according to RECIST 1.1) or death from any cause.
DCR | max 6 months
  The percentage of subjects with CR+PR+SD and last more than 4 weeks in all of the participants with measurable lesions.
OS | approximately 3 years
  Time to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China